CLINICAL TRIAL: NCT01742325
Title: The Effect of Walking Intervention on Sleep Related Symptom Distress in Pediatric Oncology Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Associate Professor, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 200904018R
Record Dates: First submitted 2012-01-31; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Childhood Cancer
Keywords: fatigue; walking; childhood cancer; sleep disturbance
MeSH Terms: conditions — Neoplasms; Fatigue; Parasomnias | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Other): To test an intervention program (two 20-minute sessions of walking around the nurse's station daily, five days a cycle) to reduce the symptoms of fatigue and pain and increase quality of sleep.
  Interventions: Behavioral: walking

INTERVENTIONS:
Behavioral: walking — two 20-minute sessions of walking around the nurse's station daily, five days a cycle
  Other Names: The effect of walking intervention on sleep related symptom

SUMMARY:
Specific aims:

Control group(2010/1~2011/6)： Aim 1: Describe the patterns of "fatigue, sleep disturbance, and pain" in children with cancer from perspectives of children and their parents over the course of one cycle (five days) of inpatient chemotherapy (CXT).

Aim 2: Determine, at various time points (during they are hospitalization various four times), the associations between fatigue, sleep disturbance, and pain over the course of four cycles (there are five days in each cycle) of CTX in children with cancer.

Aim 3: Examine the associations between a symptom cluster of fatigue, sleep disturbance, pain, child reported Quality of Life for Children with Cancer (QOLCC), parent reported uncertainty and QOL, and biomarkers over the course of four cycles of CXT in children with cancer.

Intervention group(2011/7~2012/12)： Aim 4: To test an intervention program (two 20-minute sessions of walking around the nurse's station daily, five days a cycle) to reduce the symptoms of fatigue and pain and increase quality of sleep.

DETAILED DESCRIPTION:
※ Background & Significance: Symptom management is a major issue for pediatric oncology patients and their parents. In clinical practice patients undergoing cancer treatment seldom present with a single symptom, but usually suffer from multiple symptoms simultaneously. However, when discussing symptom distress in children with cancer, studies have mostly focused on one (single) symptom. Fatigue and pain are two of the most frequent symptoms generated by cancer treatment and they attribute this to their altered sleep pattern. The new concept of the clustering of fatigue, sleep and pain needs additional research to strengthen this beginning scientific base. At this point limited empirical studies have provided evidence or foundational knowledge of the symptom clusters experienced by children with cancer, thus this is a new area and knowledge should be developed as soon as possible for management. Innovative interventions aimed at improving their physical functions such as sleep, fatigue, and pain and adherence to positive health behaviors such as regular walking are warranted. In addition, one parent of eligible children newly diagnosed with cancer will be recruited to examine their quality of life and perception of uncertainty in illness.

※ Specific aims: Control group(2010/1~2011/6)： Aim 1: Describe the patterns of "fatigue, sleep disturbance, and pain" in children with cancer from perspectives of children and their parents over the course of one cycle (five days) of inpatient chemotherapy (CXT).

Aim 2: Determine, at various time points(during they are hospitalization various four times), the associations between fatigue, sleep disturbance, and pain over the course of four cycles (there are five days in each cycle) of CTX in children with cancer.

Aim 3: Examine the associations between a symptom cluster of fatigue, sleep disturbance, pain, child reported Quality of Life for Children with Cancer (QOLCC), parent reported uncertainty and QOL, and biomarkers over the course of four cycles of CXT in children with cancer.

Intervention group(2011/7~2012/12)： Aim 4: To test an intervention program (two 20-minute sessions of walking around the nurse's station daily, five days a cycle) to reduce the symptoms of fatigue and pain and increase quality of sleep.

※ Research Design and Methods: The Human Response Model serves as a theoretical framework to guide current proposed study. The "Individual Factors" in this study includes age, gender, and type of chemotherapeutic agent patients receive as non-modifiable person factors. The "Environmental factors" includes the type of room such as single room and two beds or three beds in a room and number of other person in the room during patients stay in the hospital. The "Human responses" (during five days of CTX) includes responses of 1) physiologic such as hemoglobin, hematocrit, and urine 8-OHdG, 2) experiential such as the feelings of fatigue and pain, and 3) behavioral such as the sleep responses including sleep duration and nighttime awakenings.

Children will be eligible for this study if they (1) are aged 10 to 18 years, (2) diagnosed with cancer, (3) prescribed CTX, (4) are not receiving concomitant radiation, and (5) have not undergone bone marrow transplantation. Patients with central nervous system tumors will be ineligible because sleep problems have been associated with brain injury. Besides, patients with osteosarcoma and bone metastasis will not be recruited because they may have troubles with walking. Based on the power analysis, a total of 160 eligible patients will be recruited, N = 80 for the control and N = 80 for the intervention group.

There are a total of four observation periods (during they are hospitalization various four times)(there are five days in each period ) (O) for each diagnosed child with cancer , during next four consecutive hospitalizations for chemotherapy. The data from this study will be used to analyze the trend of symptom changes and will be as the control group. 2011/7~2012/12, an intervention (X) of two 20-minute walking will be implemented into their daily activity, one in the morning and the other one in the afternoon. Then four observation periods with the same procedures, frequency, and other described measures will be used to collect data.

Following parental consent and child assent, children will wear a wrist actigraph to monitor sleep activity every day (during they are hospitalization various four times)(there are five days in each period )and be asked to complete the Taiwanese versions of the Memorial System Assessment Scale (MSAS, 10-18), Fatigue Scale (7-12, 13-18), and the QOLCC at day 1. Then the measurements will be repeated every other day for the following consecutive five days during each cycle of CXT for at least four cycles of inpatient CTX. Parents will be asked to complete the SF-36 for their quality of life and Parent Perception Uncertainty in Illness Scale at day 0 and every other day following consecutive five days during one cycle of CXT for at least four cycles of inpatient CTX.

Descriptive time series plots of sleep variables will be generated for individual and group data. Repeated ANOVA (mixed model analysis) measurement will evaluate changes/differences in the longitudinal data relating to sleep and fatigue. Individual time-series plots will compare sleep, symptom clusters and fatigue.

※ Anticipated Results: Knowledge developed in this study can provide a starting point from which quality of life for children with cancer can be promoted through identification of factors contributing to altered sleep in hospital and the development of interventions to improve sleep.

ELIGIBILITY:
Inclusion Criteria:

* are aged 10 to 18 years
* diagnosed with cancer
* prescribed CTX
* are not receiving concomitant radiation
* have not undergone bone marrow transplantation.

Exclusion Criteria:

* patients with central nervous system tumors will be ineligible because sleep problems have been associated with brain injury.
* besides, patients with osteosarcoma and bone metastasis will not be recruited because they may have troubles with walking.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | During subjects are hospitalization various four times, and there are five days in each period
  The investigators measure the outcome by actigraph and questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ling Lee, RN,DNSc, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan